CLINICAL TRIAL: NCT06304194
Title: Pilot Study to Assess the Feasibility of Centralizing Biological Samples at Onset and Relapse of Patients Referred to CROP Centers for Molecular Characterization of Oncohematologic Pathology
Brief Title: Molecular Characterizazion and Biological Samples Centralisation of Patients Affected by Oncoematolofic Pathology
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Meyer Children's Hospital IRCCS (Other)
Responsible Party: Principal Investigator, Marinella Veltroni, Principal Investigator, Meyer Children's Hospital IRCCS
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Screening
Other Study IDs: BIOMARC_ONCO
Record Dates: First submitted 2024-02-23; First posted 2024-03-12 (Actual); Last update posted 2024-03-12 (Actual); Status verified 2024-03

CONDITIONS: Oncologic Disease; Hematologic Diseases
MeSH Terms: conditions — Hematologic Diseases

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Patients with suspected diagnostic onco-hematologic/immunologic disease (Other): All patients with suspected diagnostic onco-hematologic, onco-immunologic, and hematologic disease at onset or relapse.
  Patients undergo several procedures to complete the diagnostic process and eventually the staging of the disease
  Interventions: Other: Analysis of biological samples

INTERVENTIONS:
Other: Analysis of biological samples — The collected biological sample will be isolated and the specific nucleic acid (DNA/RNA/cfDNA) extracted for molecular analysis for understanding the reproducibility of the analysis and thus the feasibility of centralization:
  * hot spot on DNa (ddPCR/Sanger)
  * fusion genes on RNA (target resequencing)
  * Known mutation analysis by liquid biopsy (cfDNA) for somatic mutations with a mutation frequency of less than 10%
  * Tumor type-associated gene sequence analysis by Sanger sequencing and NGS

SUMMARY:
Currently, the molecular characterization of onco-hematological, onco-immunological and hematological diseases, at onset or in relapse, of patients with suspected diagnosis afferent to the CROP centers, is done through centralization of biological samples at reference laboratories outside the Tuscany Region.

In order to preserve the wealth of clinical and biological data and use it for the benefit of present and future patients treated at the CROP centers, it is useful to evaluate the feasibility of centralization and molecular typing of mutations present in tumor tissue at the IRCCS AOU Meyer Oncohematology Laboratories and subsequently the analysis of clinical data from patients with diseases not under study to lay the foundations of a translational database that can then be associated with a biobank in the future.

This will enable a targeted contribution to pediatric oncohematology research, investing in possible targeted therapies with those patient subgroups that benefit from personalized disease assessment in mind. The goal of the project is to improve the regional infrastructure dedicated to organized data collection and management of biological samples in adequate time resulting in better and more comprehensive data collection.

ELIGIBILITY:
Inclusion Criteria:

* Diagnostic suspicion of oncologic, hematologic or onco-immunologic disease
* Suspected recurrence of oncological, onco-hematological, hematological or onco -immunological disease
* Availability of biological material
* Signature of informed consent
* Age between 0 and 30 years

Exclusion Criteria:

* Failure to sign the consent
* Insufficiency of biological material for analysis
* Patients with HIV, HCV and HBV seropositivity (HBSAg) due to biohazard and bias related to patients' immunological status that could influence gene expression and tumor behavior.

Ages: 0 Years to 30 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 340 (Estimated)
Dates: Start 2023-07-05 (Actual); Primary Completion 2027-07-05 (Estimated); Study Completion 2028-07-05 (Estimated)

PRIMARY OUTCOMES:
Average sample delivery time and % of accepted sample | After 5 year from the beginning of the study
  average sample delivery time and % of samples accepted within 48 ±12 hours of collection out of total samples sent
Appropriateness sample labelling | After 5 year from the beginning of the study
  % samples correctly labelled according to IATA criteria out of total samples accepted within 48 hours
Percentage of sample suitable for RNA extraction | After 5 year from the beginning of the study
  % samples suitable for RNA extraction out of total samples intended for RNA analysis
Quantity and quality of extracted material. | After 5 year from the beginning of the study
  % of samples valid for analysis in terms of quantity of extracted material (25 ng/ul for cfDNA, 25 ng per amplicon for genomic DNA, 100 ng tot for NGS) and quality, assessed as A260/280 ratio analysis (1.8-2 per DNA).
Research report production time | After 5 year from the beginning of the study
  research report production time (from 2 weeks for known mutation analysis to 6 months for NGS).

SECONDARY OUTCOMES:
Genetic variants | After 5 year from the beginning of the study
  % variants validated with NGS and Sanger or in two independent experiments out of the total number of variants identified
Completed patient cards | After 5 year from the beginning of the study
  % of completed patient cards out of total patient cards of registered patients

CONTACTS AND LOCATIONS:
Overall Officials: Marinella Veltroni, Principal Investigator — Meyer Children's Hospital IRCCS
Locations (3):
- Italy (3):
  - Meyer Children's Hospital IRCCS, Florence
  - Azienda Ospedaliero-Universitaria Pisana, Pisa
  - Azienda Ospedaliero-Universitaria Senese, Siena